CLINICAL TRIAL: NCT02108392
Title: Characterization of Patients With Pseudoxanthoma Elasticum
Brief Title: Characterization of Pseudoxanthoma Elasticum
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Peter Charbel Issa, MD, University Hospital, Bonn
Other Study IDs: pending
Record Dates: First submitted 2014-04-01; First posted 2014-04-09 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Pseudoxanthoma Elasticum
Keywords: PXE; phenotype; eye; biomarkers
MeSH Terms: conditions — Pseudoxanthoma Elasticum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Pseudoxanthoma elasticum (PXE) is a rare multisystem disorder of autosomal recessive inheritance (OMIM# 264800) and an estimated prevalence between 1:25.000 and 1:100.000. PXE is characterized by calcification and fragmentation of connective tissue rich in elastic fibers. Due to its high content of elastic fibers, Bruch Membrane in eyes of patients affected by PXE becomes thickened and calcified. The ocular phenotype is characterized by angioid streaks and peau d'orange but also choroidal neovascularizations and chorioretinal atrophy thereby in part mimicking the phenotype of age-related macular degeneration. The disease is due to mutations of the ABCC6-gene coding for a transmembrane protein which is mainly expressed in the liver and kidney. It is hypothesized that ABCC6 is involved in the excretion of a yet unknown factor from the liver which inhibits systemic calcification. In animal models several candidates for this factor have been identified but direct evidence for such a factor in patients with PXE is still missing. The primary purpose of this study is to further investigate the ocular phenotype of patients with PXE using multimodal imaging and functional testing to delineate the impact of Bruch membrane pathology on the eye. Furthermore, possible systemic anti-calcification factors, as well as associations with the vascular alterations are investigated to gain more insights into the pathogenesis of PXE..

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Pseudoxanthoma elastcium based on histopathologic and/or genetic testing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pseudoxanthoma elasticum
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Ocular phenotype | patients will be followed longitudinally with an expected 1-year average interval between visits
  Patients are investigated using a multimodal imaging approach and visual function testing.

SECONDARY OUTCOMES:
Biomarkers in PXE | 1 day (first visit)
  Potential systemic biomarkers are investigated by collecting blood samples of PXE patients

CONTACTS AND LOCATIONS:
Overall Officials: Peter Charbel Issa, MD, Principal Investigator — Department of Ophthalmology, University of Bonn
Locations (1):
- Department of Ophthalmology, University of Bonn, Bonn, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Gliem M, Zaeytijd JD, Finger RP, Holz FG, Leroy BP, Charbel Issa P. An update on the ocular phenotype in patients with pseudoxanthoma elasticum. Front Genet. 2013 Apr 4;4:14. doi: 10.3389/fgene.2013.00014. eCollection 2013. PMID 23577018
- [Background] Finger RP, Fenwick E, Marella M, Charbel Issa P, Scholl HP, Holz FG, Lamoureux EL. The relative impact of vision impairment and cardiovascular disease on quality of life: the example of pseudoxanthoma elasticum. Health Qual Life Outcomes. 2011 Dec 12;9:113. doi: 10.1186/1477-7525-9-113. PMID 22152229
- [Background] Charbel Issa P, Finger RP, Gotting C, Hendig D, Holz FG, Scholl HP. Centrifugal fundus abnormalities in pseudoxanthoma elasticum. Ophthalmology. 2010 Jul;117(7):1406-14. doi: 10.1016/j.ophtha.2009.11.008. Epub 2010 Mar 1. PMID 20189652
- [Background] Finger RP, Charbel Issa P, Ladewig M, Gotting C, Holz FG, Scholl HP. Fundus autofluorescence in Pseudoxanthoma elasticum. Retina. 2009 Nov-Dec;29(10):1496-505. doi: 10.1097/IAE.0b013e3181aade47. PMID 19823106
- [Background] Charbel Issa P, Finger RP, Holz FG, Scholl HP. Multimodal imaging including spectral domain OCT and confocal near infrared reflectance for characterization of outer retinal pathology in pseudoxanthoma elasticum. Invest Ophthalmol Vis Sci. 2009 Dec;50(12):5913-8. doi: 10.1167/iovs.09-3541. Epub 2009 Jun 24. PMID 19553619
- [Background] Gliem M, Finger RP, Fimmers R, Brinkmann CK, Holz FG, Charbel Issa P. Treatment of choroidal neovascularization due to angioid streaks: a comprehensive review. Retina. 2013 Jul-Aug;33(7):1300-14. doi: 10.1097/IAE.0b013e3182914d2b. PMID 23719398
- [Background] Gliem M, Fimmers R, Muller PL, Brinkmann CK, Finger RP, Hendig D, Holz FG, Charbel Issa P. Choroidal changes associated with Bruch membrane pathology in pseudoxanthoma elasticum. Am J Ophthalmol. 2014 Jul;158(1):198-207.e3. doi: 10.1016/j.ajo.2014.04.005. Epub 2014 Apr 13. PMID 24727260
- [Background] Charbel Issa P, Gliem M, Holz FG, Knabbe C, Hendig D. [Pseudodominant inheritance of pseudoxanthoma elasticum]. Ophthalmologe. 2015 Aug;112(8):686-90. doi: 10.1007/s00347-014-3231-9. German. PMID 25735631
- [Background] Gliem M, Hendig D, Finger RP, Holz FG, Charbel Issa P. Reticular pseudodrusen associated with a diseased bruch membrane in pseudoxanthoma elasticum. JAMA Ophthalmol. 2015 May;133(5):581-8. doi: 10.1001/jamaophthalmol.2015.117. PMID 25764262
- [Background] Gliem M, Muller PL, Birtel J, Hendig D, Holz FG, Charbel Issa P. Frequency, Phenotypic Characteristics and Progression of Atrophy Associated With a Diseased Bruch's Membrane in Pseudoxanthoma Elasticum. Invest Ophthalmol Vis Sci. 2016 Jun 1;57(7):3323-30. doi: 10.1167/iovs.16-19388. PMID 27367499
- [Background] Gliem M, Muller PL, Birtel J, McGuinness MB, Finger RP, Herrmann P, Hendig D, Holz FG, Charbel Issa P. Quantitative Fundus Autofluorescence in Pseudoxanthoma Elasticum. Invest Ophthalmol Vis Sci. 2017 Dec 1;58(14):6159-6165. doi: 10.1167/iovs.17-22007. PMID 29214314
- See also: Webpage of the University Eye Hospital of Bonn — http://www.augenklinik.uni-bonn.de/